CLINICAL TRIAL: NCT02844543
Title: EYE-TRAC Advance: Technology Verification (ETA-TV) Cohort 1
Acronym: ETA-TV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Brain Trauma Foundation (Other); United States Department of Defense (U.S. Federal Agency); Food and Drug Administration (FDA) (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamshid Ghajar, Clinical Professor of Neurosurgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 34662
Record Dates: First submitted 2016-06-30; First posted 2016-07-26 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Eye-tracking
Keywords: concussion, eye-tracking, athletes, vision
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Athletes (Experimental): Participants will be evaluated using the EYE-SYNC eye-tracking device, Desktop Eye-Tracker, and Sport Concussion Assessment Tool (SCAT-3) tool.
  Interventions: Device: EYE-SYNC eye-tracking device; Other: SCAT-3; Device: Desktop Eye-Tracker

INTERVENTIONS:
Device: EYE-SYNC eye-tracking device — The EYE-SYNC® portable eye-tracking system. The eye tracker is a handheld isolated display environment with embedded eye tracking sensors. The eye tracker is connected to a high-performance Windows tablet though a customized docking station. Included accessories with EYE-SYNC are a U.S. tablet power supply adapter and disposable sanitary masks. Participants are asked to follow a dot with their eyes, as the dot moves on the screen of the EYE-SYNC device.
Other: SCAT-3 — The Symptom subtest of SCAT-3 assessment tool will be administered to participants.
Device: Desktop Eye-Tracker — Eye movements are recorded with an eye tracking system (Desktop Eye-Tracker, Eyelink CR, SR Research) with up to 1000 Hz temporal resolution. The target stimulus is presented on a computer screen approximately 50 cm from the participant. Participants are asked to follow a dot with their eyes, as the dot moves on the monitor screen of the desk-top eye-tracking device.

SUMMARY:
This study will assess the effects of exercise and non-concussive bodily contact on eye-tracking scores collected by the EYE-SYNC eye-tracking device.

DETAILED DESCRIPTION:
The investigators propose to prospectively study a cohort of 18-25-year-old athletes. Athletes will be tested with the EYE-SYNC eye-tracking device prior to the start of an athletic practice or competition (pre-test) and then after the conclusion of the practice/competition (post-test). The investigators hope to understand if eye-tracking scores are effected by exercise and non-concussive bodily contact commonly incurred during athletic play.

ELIGIBILITY:
Inclusion criteria

* Athletes between the age of 18- 25-years-old.
* 20/30 or better eyesight (corrected vision allowed).
* English fluency.

Exclusion criteria

Note: Under Cohort 1, Athletes that have conditions listed below will not be excluded from the study. They will be enrolled and their subject data will be analyzed separately from subjects who do not endorse any significant medical hx under neurological, eye-sight, or psychiatric categories.

* Clinical diagnosis of a neurological condition including the following: Stroke, Multiple Sclerosis, Epilepsy, Brain Tumor/Cancer, Nystagmus and/or other major neurological condition.
* Clinical diagnosis of any of the following eye-sight abnormalities: Uncorrected Amblyopia, Uncorrected Myopia, Uncorrected Presbyopia, Uncorrected Farsightedness, or Uncorrected Astigmatism.
* Psychiatric history with any of the following:

  1. Clinical diagnosis of a psychotic disorder, bipolar disorder - lifetime
  2. Clinical diagnosis of ADHD or ADD - Lifetime
  3. Clinical diagnosis of major depressive disorder - within last year
  4. Clinical diagnosis of substance abuse disorder - within last year
  5. Clinical diagnosis of major anxiety disorder - within last year

     MEDICATION
  6. Requires use of a psychotropic medication.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Little, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Athletes: Participants were tested with the EYE-SYNC eye-tracking device, the Desktop Eye-tracker, and SCAT-3 Symptom subtest.
Period: Overall Study
Arm/Group | Athletes
Started | 155
Completed | 150
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Did not meet eligibility criteria | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol were included in the analysis.
Arm/Group | Athletes
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Eye-tracking Score Before and After Practice or Game: Phase Error
Description: The EYE-SYNC test was performed before and after practice to analyze the effect of exercise and sub-concussive impact. The movement of eye was tracked using EYE-SYNC. The data were recorded in a surface tablet connected to EYE-SYNC.
  Phase error is defined as the difference in degrees between movement of the target and the movement of the eye. Positive values indicate the eye is ahead of the target; negative values indicate the eye is behind the target.
Time Frame: Up to 6 hours
Population: Participants with evaluable data at the respective time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Athletes
Number analyzed (Participants) | 155
Degrees
  Prior to practice/game: number analyzed (Participants) | 150
  Prior to practice/game | -0.6 (4.0)
  After practice/game: number analyzed (Participants) | 136
  After practice/game | -0.8 (0.5)

2. Secondary Outcome: Changes in Sport Concussion Assessment Tool (SCAT-3) Standardized Assessment of Concussion (SAC) Score
Description: Change in SCAT-3 SAC score before and after practice or game is reported. The SAC score is based on the following assessments: number of symptoms (22 points), symptom severity (132 points), orientation (5 points), immediate memory (15 points), concentration (5 points), and delayed recall (5 points). Scores are summed for a possible range of 0 to 184, with lower scores corresponding to fewer concussion symptoms, and higher scores corresponding to more concussion symptoms.
Time Frame: Day of study/event (up to 6 hours)
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Athletes
Number analyzed (Participants) | 150
units on a scale | -0.6 (3.6)

3. Primary Outcome: Changes in the Eye-tracking Score Before and After Practice or Game: Tangential and Radial Error
Description: The EYE-SYNC test was performed before and after practice to analyze the effect of exercise and sub-concussive impact. The movement of eye was tracked using EYE-SYNC. The data were recorded in a surface tablet connected to EYE-SYNC.
  Tangential and radial error are defined as degrees of variation in eye tracking along a circular path (tangential) and at 90 degrees to the tangential path (radial). Positive values indicate the eye is ahead of the target; negative values indicate the eye is behind the target.
Time Frame: Up to 6 hours
Population: Participants with evaluable data at the respective time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: Degrees of variation
Arm/Group | Athletes
Number analyzed (Participants) | 155
Degrees of variation
  Tangential: prior to practice/game: number analyzed (Participants) | 150
  Tangential: prior to practice/game | 1.2 (0.8)
  Tangential: after practice/game: number analyzed (Participants) | 136
  Tangential: after practice/game | 1.1 (0.7)
  Radial: prior to practice/game: number analyzed (Participants) | 134
  Radial: prior to practice/game | 0.9 (0.4)
  Radial: after practice/game: number analyzed (Participants) | 136
  Radial: after practice/game | 0.8 (0.5)

4. Primary Outcome: Changes in the Eye-tracking Score Before and After Practice or Game: Vertical and Horizontal Gain
Description: The EYE-SYNC test was performed before and after practice to analyze the effect of exercise and sub-concussive impact. The movement of eye was tracked using EYE-SYNC. The data were recorded in a surface tablet connected to EYE-SYNC.
  Vertical and horizontal gain are defined as the ratio of velocity (velocity of the eye:velocity of the target). Positive values indicate the eye is ahead of the target; negative values indicate the eye is behind the target.
Time Frame: Up to 6 hours
Population: Participants with evaluable data at the respective time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: Ratio of velocity (degrees per second)
Arm/Group | Athletes
Number analyzed (Participants) | 155
Ratio of velocity (degrees per second)
  Horizontal: prior to practice/game: number analyzed (Participants) | 150
  Horizontal: prior to practice/game | 0.9 (0.1)
  Horizontal: after practice/game: number analyzed (Participants) | 136
  Horizontal: after practice/game | 0.9 (0.1)
  Vertical: prior to practice/game: number analyzed (Participants) | 134
  Vertical: prior to practice/game | 0.8 (0.1)
  Vertical: after practice/game: number analyzed (Participants) | 136
  Vertical: after practice/game | 0.8 (0.1)

ADVERSE EVENTS:
Time Frame: Day of study/event (up to 6 hours)
Arm/Group | Athletes
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes